CLINICAL TRIAL: NCT06064825
Title: Long Term Follow-up of the TREOCAPA (Prophylactic TREatment Of the duCtus Arteriosus in Preterm Infants by Acetaminophen) Study (TREOCAPA-LT)
Brief Title: Long Term Follow-up of the TREOCAPA Study (TREOCAPA-LT)
Acronym: TREOCAPA-LT
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C23-31; 2023-A01418-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-09-15; First posted 2023-10-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Patency of the Ductus Arteriosus Acetaminophen Extreme Prematurity
Keywords: Premature infants; persistent ductus arteriosus; paracetamol/acetaminophen; long term outcome
MeSH Terms: conditions — Premature Birth; Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients received the investigational medicinal product acetaminophen in their first 5 days of life: This group of patients received the investigational product in their first 5 days of life during the Treocapa trial
  Interventions: Other: 2 year follow-up of neurodevelopment using a parental questionnaire
- patients received the placebo (NaCl) in their first 5 days of life: This group of patients received the placebo in their first 5 days of life during the Treocapa trial
  Interventions: Other: 2 year follow-up of neurodevelopment using a parental questionnaire

INTERVENTIONS:
Other: 2 year follow-up of neurodevelopment using a parental questionnaire — A parental questionnaire, using the PARCA-R instrument, is given to measure cognitive outcome at 2 years of corrected age for children included in the Treocapa Trial

SUMMARY:
The ductus arteriosus (DA) is a large channel connecting the main pulmonary trunk with the descending aorta. In extremely preterm infants, the DA frequently fails to close and this results in a condition called patent ductus arteriosus (PDA). In these patients, PDA has been associated with increased mortality and morbidity in the neonatal period, and neonatal morbidities may in turn be associated with later deficits in cognitive functioning. PDA treatment with COX inhibitors, as ibuprofen or indomethacin, aiming at closing the PDA have been associated with numerous adverse effects and failed to demonstrate significant clinical benefits. Early treatment of PDA with paracetamol (acetaminophen ) has been proposed as an alternative to COX inhibitors. The ongoing pan-European TREOCAPA phase III study (NCT04459117) is a multicentre, double-blind, randomised, placebo-controlled superiority trial that assesses prophylactic use of paracetamol to improve survival without severe neonatal morbidity until discharge from hospital in infants of 23-28 weeks of gestational age. As long-term follow-up was not planned by the TREOCAPA protocol, TREOCAPA-LT study will use an existing European research infrastructure, the RECAP Preterm platform (https://recap-preterm.eu/), to follow-up the patients enrolled in the TREOCAPA trial using a parent-report questionnaire at 2 years of corrected age.

The TREOCAPA-LT primary hypothesis is that there will be improved cognitive outcome at 2 years of corrected age in children born at less than 29 weeks of gestational age who were treated with paracetamol during the first 5 days of life in the TREOCAPA phase III trial.

DETAILED DESCRIPTION:
The ductus arteriosus (DA) is a large channel found normally in all mammalian foetuses, connecting the main pulmonary trunk with the left-sided descending aorta. During fetal life, it diverts most of the combined ventricular output away from the lungs toward the placenta. In full-term newborns, the DA is functionally open in all newborns and its constriction and closure, within 24 to 48 hours after delivery, are part of the normal process of postnatal adaptation. In extremely preterm infants, ie, those born before 29 weeks of gestation, the DA frequently fails to close and this results in a condition called patent ductus arteriosus (PDA). In these patients, PDA has been associated with increased mortality and morbidity in the neonatal period, and neonatal morbidities may in turn be associated with later deficits in cognitive functioning. Inhibition of prostaglandin synthesis, through inhibition of the cyclo-oxygenase (COX) enzymes, results in ductal constriction. However, treatments with COX inhibitors, as ibuprofen or indomethacin, aiming at closing the PDA have been associated with numerous adverse effects and failed to demonstrate significant clinical benefits. Prophylactic use of indomethacin or ibuprofen has been shown to reduce subsequent development of PDA but not to reduce mortality or morbidity. Further, investigations of early cardiac ultrasound-targeted treatment of a large PDA using indomethacin and ibuprofen do not show efficacy on primary outcomes of neonatal death or morbidity. Although this evidence base shows that prophylactic treatment by indomethacin or ibuprofen cannot be recommended, evidence from observational studies suggests that early (during the first 3 days of life) conservative treatment should not be recommended either. Two observational studies indicated that ignoring a PDA during the first days of life is associated with increase in mortality or morbidity. Our interpretation of these results is that screening echocardiography of large ductus arteriosus and early targeted treatment using echocardiography reduce pulmonary haemorrhage, but that the use of drugs with severe adverse effects may cancel expected beneficial effects on the occurrence of death or morbidity.

The use of a medication with an effect on PDA and that has fewer adverse effects is therefore desirable. Early treatment of PDA with paracetamol (acetaminophen) has been proposed as an alternative to COX inhibitors. According to a recent meta-analysis, use of paracetamol has a comparable effectiveness to close a PDA, and fewer harmful effects. However, only few extremely preterm infants were included in this meta-analysis. Therefore, efficacy and safety of paracetamol for PDA treatment in this population required further studies.

The ongoing pan-European TREOCAPA phase III study (NCT04459117) is a multicentre, double-blind, randomised, placebo-controlled superiority trial that assesses prophylactic use of paracetamol to improve survival without severe neonatal morbidity until discharge from hospital in infants of 23-28 weeks of gestational age.12 The trial has been powered to identify an absolute difference of 10% in the primary outcome, survival without severe neonatal morbidity (defined as any of: bronchopulmonary dysplasia grade 3 according to National Institute of Health criteria, necrotising enterocolitis stage 2 or 3 using Bell's criteria, intraventricular haemorrhage grade III or IV using the classification of Papile et al, or any evidence of cystic periventricular leukomalacia), corresponding to an increase from 50% to 60% in the rate between groups at hospital discharge. It aims to recruit 398 infants born at 27-28 weeks of gestation, and 396 infants born at 23-26 weeks of gestation. The first patients were recruited in October 2020 and the recruitment period is anticipated to last until April 2024 at the latest.

The TREOCAPA phase III trial is ambitious and innovative in its scope, including more than 40 hospitals in 16 countries. However, long-term follow-up was not included in the TREOCAPA protocol. The follow-up of infants enrolled in clinical trials enables to measure the long-term effectiveness and safety of interventions performed in the neonatal period. In particular for exposition to paracetamol in the neonatal period, data from randomized studies are very limited, while long-term adverse effects of paracetamol, including notably behavioral problems, have been raised. There is hence a need to understand longer term outcomes for the infants enrolled in this study, as these longer-term endpoints correspond to important patient-valued outcomes and are critical to determining the comparative effectiveness of interventions. The working hypothesis, if the intervention has a positive impact on short-term endpoints, is that longer term outcomes will be better in the intervention group, reflecting reduced morbidity at discharge home from the neonatal hospitalisation.

As long-term follow-up was not planned by the TREOCAPA phase III protocol, TREOCAPA-LT study will use an existing European research infrastructure, the RECAP Preterm platform to follow-up patients enrolled in the TREOCAPA cohort at 2 years of corrected age. This platform federates 23 European longitudinal observational cohorts of children born very preterm. The platform includes expertise, tools and infrastructure to follow patients enrolled in trials. By integrating trial follow-up in this platform, it is also possible to compare patients enrolled in the TREOCAPA trial with those from population-based samples, allowing assessment of transportability of trial results.

Follow-up at 2 years of age is recommended as the focus for the first phase of long-term outcome monitoring and has become the de facto age which is used in many published and ongoing clinical trials. Furthermore, many hospital services provide follow-up for their patients until at least 2 years of age, and research contact with the families at this point provides an opportunity to maintain contact and demonstrate to patients the ongoing importance of their involvement in the study.

The TREOCAPA-LT primary hypothesis is that there will be improved cognitive outcome at 2 years of corrected age in children born at less than 29 weeks of gestational age who were treated with paracetamol during the first 5 days of life in the TREOCAPA trial.

Secondary hypotheses are that, among children treated with paracetamol/acetaminophen during the first 5 days of life:

1. There will be reduced moderate or severe neurodevelopmental impairment, defined as the presence of at least one of the following: PARCA-R non-verbal cognitive score less than two standard deviations below the mean (score <70) moderate-severe motor impairment, unilateral or bilateral deafness or blindness.
2. There will be reduced need for secondary hospitalisations following the initial neonatal hospitalisation.
3. There will be reduced long term health care utilisation costs associated with extremely preterm birth.

Secondary hypotheses also relate to the use of the RECAP Preterm platform of observational VPT cohorts in this study. These are that:

1. As a trial population, the children born VPT included in the TREOCAPA-LT study will differ from those included in population-based observational cohorts in their perinatal characteristics and possibly in their health and developmental outcomes.
2. That these differences in population characteristics can affect the transportability of the trial results to other populations of VPT infants.

ELIGIBILITY:
Inclusion Criteria:

* were included in the TREOCAPA phase III RCT in participating centres
* are aged between 23.5 and 27.5 months corrected age during the study period

Exclusion Criteria:

* if the local investigator does not have up-to-date contact information allowing contact with parents
* if the child's vital status cannot be ascertained
* if the child is nearing the end of his life or experiencing a severe medical event as assessed by the local investigator
* if the child has become subject to a legal protection measure preventing their ongoing participation in clinical research
* if either parent or guardian opts out of participating
* language barrier

Ages: 23 Months to 27 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population for the follow-up study of the TREOCAPA trial consists of all children included in phase III of the trial from centres participating in the follow-up study. The parents of children who survived to two years corrected age and meet the criteria for inclusion will be offered the opportunity to complete the questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Non-verbal cognition at 2 years corrected age | from 23,5 to 27,5 months of corrected age
  Non-verbal cognitive (NVC) scale score from the Parent Report of Children's Abilities-Revised (PARCA-R) questionnaire, administered using an on-line parental questionnaire. The score is standardised such that it has a mean of 100 and a standard deviation of 15. Lower scores mean worse outcomes.

SECONDARY OUTCOMES:
Survival without moderate or severe cognitive impairment | from 23,5 to 27,5 months of corrected age
  Definied as survival to 2 years corrected age with a PARCA-R NVC scale score less than 2 standard deviations below the mean.
Survival without moderate or severe neurodevelopmental impairment based on the presence of at least one of the impairments in the description : | from 23,5 to 27,5 months of corrected age
  1. the PARCA-R NVC < 2 standard deviations below the mean;
  2. moderate to severe motor impairment, as measured using parent reported questions, defined as a child unable to: walk without assistance or aids or sit or hold their head up without support19;
  3. unilateral or bilateral deafness or blindness as measured by parent reported questions: if the child is deaf or has functional hearing loss requiring correction with aids but still has difficulty hearing, or if the child is blind or able to see light only19.
Health service use and costs | from 23,5 to 27,5 months of corrected age
  Reported by parents in the questionnaire, using questions on visits to health service providers and other costs associated with care of the children that have been used in previous European studies

OTHER OUTCOMES:
Comparisons of the results with observational cohorts of very preterm infants for maternal sociodemographic characteristics | This analysis will be carried during the 12 months after the end of data collection.
  Descriptive statistics on maternal sociodemographic characteristics
Comparisons of the results with observational cohorts of very preterm infants for gestational age | This analysis will be carried during the 12 months after the end of data collection.
  Descriptive statistics on gestational age
Comparisons of the results with observational cohorts of very preterm infants on sex | This analysis will be carried during the 12 months after the end of data collection.
  Descriptive statistics on sex
Comparisons of the results with observational cohorts of very preterm infants for complication of pregnancy | This analysis will be carried during the 12 months after the end of data collection.
  Descriptive statistics on complications of pregnancy
Comparisons of the results with observational cohorts of very preterm infants for birth | This analysis will be carried during the 12 months after the end of data collection.
  Descriptive statistics on complication of birth
Comparisons of the results with observational cohorts of very preterm infants for neonatal morbidities | This analysis will be carried during the 12 months after the end of data collection.
  Descriptive statistics on neonatal morbidities
Comparisons of the results with observational cohorts of very preterm infants for mortality | This analysis will be carried during the 12 months after the end of data collection.
  Descriptive statistics on mortality
Comparisons of the results with observational cohorts of very preterm infants for neurodevelopment | This analysis will be carried during the 12 months after the end of data collection.
  Descriptive statistics on two-year neurodevelopment

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Zeitlin, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (8):
- France (8):
  - CHU d'Angers, Angers
  - Hôpital Femme Mère Enfant, Bron
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - Cochin - APHP, Paris
  - Hopital Robert Debré, Paris
  - CHU de Strasbourg, Strasbourg
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clyman RI. Ibuprofen and patent ductus arteriosus. N Engl J Med. 2000 Sep 7;343(10):728-30. doi: 10.1056/NEJM200009073431009. No abstract available. PMID 10974138
- [Background] Hamrick SEG, Sallmon H, Rose AT, Porras D, Shelton EL, Reese J, Hansmann G. Patent Ductus Arteriosus of the Preterm Infant. Pediatrics. 2020 Nov;146(5):e20201209. doi: 10.1542/peds.2020-1209. PMID 33093140
- [Background] Mitra S, de Boode WP, Weisz DE, Shah PS. Interventions for patent ductus arteriosus (PDA) in preterm infants: an overview of Cochrane Systematic Reviews. Cochrane Database Syst Rev. 2023 Apr 11;4(4):CD013588. doi: 10.1002/14651858.CD013588.pub2. PMID 37039501
- [Background] Fowlie PW, Davis PG, McGuire W. Prophylactic intravenous indomethacin for preventing mortality and morbidity in preterm infants. Cochrane Database Syst Rev. 2010 Jul 7;2010(7):CD000174. doi: 10.1002/14651858.CD000174.pub2. PMID 20614421
- [Background] Ohlsson A, Walia R, Shah SS. Ibuprofen for the treatment of patent ductus arteriosus in preterm or low birth weight (or both) infants. Cochrane Database Syst Rev. 2018 Sep 28;9(9):CD003481. doi: 10.1002/14651858.CD003481.pub7. PMID 30264852
- [Background] Kluckow M, Jeffery M, Gill A, Evans N. A randomised placebo-controlled trial of early treatment of the patent ductus arteriosus. Arch Dis Child Fetal Neonatal Ed. 2014 Mar;99(2):F99-F104. doi: 10.1136/archdischild-2013-304695. Epub 2013 Dec 6. PMID 24317704
- [Background] Roze JC, Cambonie G, Le Thuaut A, Debillon T, Ligi I, Gascoin G, Patkai J, Beuchee A, Favrais G, Flamant C, Durrmeyer X, Clyman R. Effect of Early Targeted Treatment of Ductus Arteriosus with Ibuprofen on Survival Without Cerebral Palsy at 2 Years in Infants with Extreme Prematurity: A Randomized Clinical Trial. J Pediatr. 2021 Jun;233:33-42.e2. doi: 10.1016/j.jpeds.2020.12.008. Epub 2020 Dec 9. PMID 33307111
- [Background] Liebowitz M, Clyman RI. Prophylactic Indomethacin Compared with Delayed Conservative Management of the Patent Ductus Arteriosus in Extremely Preterm Infants: Effects on Neonatal Outcomes. J Pediatr. 2017 Aug;187:119-126.e1. doi: 10.1016/j.jpeds.2017.03.021. Epub 2017 Apr 7. PMID 28396025
- [Background] Roze JC, Cambonie G, Marchand-Martin L, Gournay V, Durrmeyer X, Durox M, Storme L, Porcher R, Ancel PY; Hemodynamic EPIPAGE 2 Study Group. Association Between Early Screening for Patent Ductus Arteriosus and In-Hospital Mortality Among Extremely Preterm Infants. JAMA. 2015 Jun 23-30;313(24):2441-8. doi: 10.1001/jama.2015.6734. PMID 26103028
- [Background] Clyman RI, Liebowitz M, Kaempf J, Erdeve O, Bulbul A, Hakansson S, Lindqvist J, Farooqi A, Katheria A, Sauberan J, Singh J, Nelson K, Wickremasinghe A, Dong L, Hassinger DC, Aucott SW, Hayashi M, Heuchan AM, Carey WA, Derrick M, Fernandez E, Sankar M, Leone T, Perez J, Serize A; PDA-TOLERATE (PDA: TO LEave it alone or Respond And Treat Early) Trial Investigators. PDA-TOLERATE Trial: An Exploratory Randomized Controlled Trial of Treatment of Moderate-to-Large Patent Ductus Arteriosus at 1 Week of Age. J Pediatr. 2019 Feb;205:41-48.e6. doi: 10.1016/j.jpeds.2018.09.012. Epub 2018 Oct 16. PMID 30340932
- [Background] Jasani B, Mitra S, Shah PS. Paracetamol (acetaminophen) for patent ductus arteriosus in preterm or low birth weight infants. Cochrane Database Syst Rev. 2022 Dec 15;12(12):CD010061. doi: 10.1002/14651858.CD010061.pub5. PMID 36519620
- [Background] Marlow N, Doyle LW, Anderson P, Johnson S, Bhatt-Mehta V, Natalucci G, Darlow BA, Davis JM, Turner MA; International Neonatal Consortium (INC). Assessment of long-term neurodevelopmental outcome following trials of medicinal products in newborn infants. Pediatr Res. 2019 Nov;86(5):567-572. doi: 10.1038/s41390-019-0526-1. Epub 2019 Aug 9. PMID 31398720
- [Background] Masarwa R, Levine H, Gorelik E, Reif S, Perlman A, Matok I. Prenatal Exposure to Acetaminophen and Risk for Attention Deficit Hyperactivity Disorder and Autistic Spectrum Disorder: A Systematic Review, Meta-Analysis, and Meta-Regression Analysis of Cohort Studies. Am J Epidemiol. 2018 Aug 1;187(8):1817-1827. doi: 10.1093/aje/kwy086. PMID 29688261
- [Background] Baker BH, Lugo-Candelas C, Wu H, Laue HE, Boivin A, Gillet V, Aw N, Rahman T, Lepage JF, Whittingstall K, Bellenger JP, Posner J, Takser L, Baccarelli AA. Association of Prenatal Acetaminophen Exposure Measured in Meconium With Risk of Attention-Deficit/Hyperactivity Disorder Mediated by Frontoparietal Network Brain Connectivity. JAMA Pediatr. 2020 Nov 1;174(11):1073-1081. doi: 10.1001/jamapediatrics.2020.3080. PMID 32986124
- [Background] Inoue K, Ritz B, Ernst A, Tseng WL, Yuan Y, Meng Q, Ramlau-Hansen CH, Strandberg-Larsen K, Arah OA, Obel C, Li J, Olsen J, Liew Z. Behavioral Problems at Age 11 Years After Prenatal and Postnatal Exposure to Acetaminophen: Parent-Reported and Self-Reported Outcomes. Am J Epidemiol. 2021 Jun 1;190(6):1009-1020. doi: 10.1093/aje/kwaa257. PMID 33230558
- [Background] Johnson S, Bountziouka V, Brocklehurst P, Linsell L, Marlow N, Wolke D, Manktelow BN. Standardisation of the Parent Report of Children's Abilities-Revised (PARCA-R): a norm-referenced assessment of cognitive and language development at age 2 years. Lancet Child Adolesc Health. 2019 Oct;3(10):705-712. doi: 10.1016/S2352-4642(19)30189-0. Epub 2019 Aug 8. PMID 31402196
- [Background] Draper ES, Zeitlin J, Manktelow BN, Piedvache A, Cuttini M, Edstedt Bonamy AK, Maier R, Koopman-Esseboom C, Gadzinowski J, Boerch K, van Reempts P, Varendi H, Johnson SJ; EPICE group. EPICE cohort: two-year neurodevelopmental outcomes after very preterm birth. Arch Dis Child Fetal Neonatal Ed. 2020 Jul;105(4):350-356. doi: 10.1136/archdischild-2019-317418. Epub 2019 Nov 5. PMID 31690558
- [Background] Seppanen AV, Bodeau-Livinec F, Boyle EM, Edstedt-Bonamy AK, Cuttini M, Toome L, Maier RF, Cloet E, Koopman-Esseboom C, Pedersen P, Gadzinowski J, Barros H, Zeitlin J; Effective Perinatal Intensive Care in Europe (EPICE) research group. Specialist health care services use in a European cohort of infants born very preterm. Dev Med Child Neurol. 2019 Jul;61(7):832-839. doi: 10.1111/dmcn.14112. Epub 2018 Dec 3. PMID 30508225
- [Background] Seppanen AV, Draper ES, Petrou S, Barros H, Aubert AM, Andronis L, Kim SW, Maier RF, Pedersen P, Gadzinowski J, Lebeer J, Aden U, Toome L, van Heijst A, Cuttini M, Zeitlin J; SHIPS Research Group. High Healthcare Use at Age 5 Years in a European Cohort of Children Born Very Preterm. J Pediatr. 2022 Apr;243:69-77.e9. doi: 10.1016/j.jpeds.2021.12.006. Epub 2021 Dec 16. PMID 34921871